CLINICAL TRIAL: NCT05731583
Title: Telemonitoraggio Domiciliare Della Saturazione Arteriosa di Ossigeno in Pazienti COVID-19
Acronym: SATCoV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4985
Record Dates: First submitted 2023-02-14; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recovering COVID: Subjects with hospitalization due to a confirmed diagnosis of Sars-CoV-2 infection, that were considered eligible for home monitoring.
  Interventions: Device: Home pulse oximetry monitoring
- Ongoing COVID: Subjects with confirmed new diagnosis of Sars-CoV-2 infection, not requiring immediate hospitalization.
  Interventions: Device: Home pulse oximetry monitoring

INTERVENTIONS:
Device: Home pulse oximetry monitoring — A digital application and a wireless oximeter were provided to both groups. Oxygen saturation, heart rate and (optional) body temperature were monitored at least twice a day.

SUMMARY:
The COVID-19 pandemic created an urgent need to implement digital health solutions for remote clinical management of infected patients who could be monitored at home. The Gemelli Polyclinic in Rome provided a digital health program (SATCOV) to monitor at home newly diagnosed COVID-19 patient, or after an early discharge from the COVID units.

A digital application and a wireless oximeter were provided to patients. Oxygen saturation, heart rate and body temperature were monitored. The aim is to evaluate the feasibility and safety of the oxygen saturation telemonitoring in COVID-19 patients.

Clinicians personalized their remote assistance defining specific alerts for each patient and/or required a timely hospitalization in a dedicated COVID unit if necessary.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age>18)
* confirmed diagnosis of Sars-CoV-2 infection by a positive nasopharyngeal and oropharyngeal swab (PCR or rapid test)
* clinical condition compatible with hospital discharge (for recoving COVID group) or home management (for ongoing COVID group)

Exclusion Criteria:

* non-autonomous patients
* patients without a smartphone and home internet connection
* patients unable to refer to emergency room in less than 2 hours or unable to observe home isolation
* the presence of severe comorbidities that could compromise the safety of telemonitoring

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients of any gender, with confirmed diagnosis of Sars-CoV-2 infection by a positive nasopharyngeal and oropharyngeal swab (PCR or rapid test)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients without missing days of telemonitoring/total patients | 14 days
  Number of patients without missing days of telemonitoring/total patients

SECONDARY OUTCOMES:
Oxygen saturation measurements | 14 days
  Number of oxygen saturation measurements performed/total measurements required by protocol
Number of subject hospitalized/total patients | 3 yars
  Number of subject hospitalized/total patients
Descriptive statistics | 14 days
  Groups' description of their clinical and demographics characteristics
Correlation between the number of comorbidities and smoking status and SpO2 nadir | 14 days
  Correlation between the number of comorbidities and smoking status and SpO2 nadir
Cost efficacy | 14 days
  Calculation of resources spent per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No